CLINICAL TRIAL: NCT05219253
Title: A Phase 3, Randomised, Observer-blind, Placebo-controlled, Multi-centre Study to Evaluate the Immune Response and Safety of the Herpes Zoster Subunit Vaccine When Administered Intramuscularly on a 2-dose Schedule in Adults Aged 50 Years and Older in India
Brief Title: A Study on the Immune Response and Safety of a Vaccine Against Herpes Zoster in Adults Aged 50 Years and Older in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 214461
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Herpes Zoster
Keywords: Shingles; Herpes Zoster subunit vaccine; Immunogenicity; Safety; Adults aged 50 years and older; India
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data was collected in an observer-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HZ/su Group (Experimental): Participants randomized to the HZ/su group received two doses of HZ/su vaccine, administered at Day 1 and Month 2.
  Interventions: Biological: HZ/su
- Placebo Group (Placebo Comparator): Participants randomized to the Placebo group received two doses of Placebo, administered at Day 1 and Month 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HZ/su — Two doses of the HZ/su vaccine administered intramuscularly, one each at Day 1 and Month 2.
  Arms: HZ/su Group
Drug: Placebo — Two doses of Placebo (lyophilised sucrose reconstituted with saline [NaCl] solution) administered intramuscularly, one each at Day 1 and Month 2.
  Arms: Placebo Group

SUMMARY:
The purpose of this study was to evaluate the humoral immunogenicity and safety of 2 doses of GSK Biologicals' Herpes Zoster subunit vaccine (HZ/su) administered for the prevention of Herpes Zoster (HZ) in adults aged 50 years of age (YOA) or older from India.

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or participant's legally acceptable representative(s) (LAR) who in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant and/or participant's LAR(s) after the study has been explained according to local regulatory requirements and prior to performance of any study-specific procedure.
* A male or female aged 50 YOA or older at the time of the first study intervention.
* Healthy participants or medically stable patients as established by medical history and clinical examination before entering into the study.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the study intervention administration series.

Exclusion Criteria:

Medical conditions

* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s) vaccine or study materials or equipment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of HZ.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.

Prior/Concomitant therapy

• Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before first dose and ending 30 days after the last dose of study intervention administration with the exception of licensed pneumococcal vaccines and non-replicating vaccines may be administered up until 8 days prior to Dose 1 and/or Dose 2 and/or at least 14 days after any dose of study intervention.

[In case an emergency mass vaccination for an unforeseen public health threat (e.g. a pandemic) is recommended and/or organised by the public health authorities, outside the routine immunisation programme, the time period described above can be reduced if necessary for that vaccine provided it is used according to local governmental recommendations and that the Sponsor is notified accordingly.]

* Planned administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study intervention up to 1 month post-dose 2 (Month 3) or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine. For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day or equivalent is not allowed. Inhaled, intra-articular and topical steroids are allowed.
* Previous vaccination against varicella or HZ.

Prior/Concurrent clinical study experience Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/ invasive medical device).

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months of last study intervention administration.
* Indications of drug abuse or excess alcohol use as deemed by investigator to potentially confound safety assessments or render participant unable or unlikely to adhere to protocol requirements.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- India (9):
  - GSK Investigational Site, Visakhapatnam, Andhra Pradesh
  - GSK Investigational Site, North Guwāhāti, Assam
  - GSK Investigational Site, Ahmedabad, Gujarat
  - GSK Investigational Site, Mumbai, Maharashtra
  - GSK Investigational Site, Chandigarh, Punjab
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Mysore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Naficy A, Chugh Y, Tariq M, Hawksworth H, Sankhe LR, Mwakingwe-Omari A. Immune response and safety of the adjuvanted recombinant zoster vaccine in adults 50 years of age and older in India: A randomized phase 3 trial. Vaccine. 2025 Mar 19;50:126819. doi: 10.1016/j.vaccine.2025.126819. Epub 2025 Feb 10. PMID 39923547
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in India.
Pre-assignment Details: All 288 participants enrolled in this study received 2 doses of the study interventions and were included in the Exposed Set. A total of 285 participants completed the study.
Groups:
- HZ/suSeq Group: Participants randomized to the HZ/su group received two doses of HZ/su vaccine, administered at Day 1 and Month 2.
Period: Overall Study
Arm/Group | HZ/suSeq Group | Placebo Group
Started | 143 | 145
Completed | 142 | 143
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HZ/suSeq Group | Placebo Group | Total
Number analyzed (Participants) | 143 | 145 | 288
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (7.2) | 58.2 (7.0) | 58.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 99 | 97 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - CENTRAL / SOUTH ASIAN HERITAGE | 140 | 141 | 281
  ASIAN - SOUTH EAST ASIAN HERITAGE | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Showing a Vaccine Response for Anti-glycoprotein E (gE)
Description: A participant with vaccine response for anti-gE was defined as a participant with:
  * at least a 4-fold greater post-last vaccination anti-gE antibody (Ab) concentration as compared to the pre-vaccination anti-gE Ab concentration, for participants who were seropositive at baseline, or
  * at least a 4-fold greater post-last vaccination anti-gE Ab concentration as compared to the anti-gE Ab cut-off value for seropositivity, for participants who were seronegative at baseline.
Time Frame: At 1 month post-Dose 2 of study intervention administration (Month 3)
Population: This analysis was performed on the Per Protocol Set, which included all eligible participants who received all doses as per protocol, complied with allowed dosing/blood draw intervals, without intercurrent conditions that may have interfered with immunogenicity, without prohibited concomitant medication/vaccination and with immunogenicity results available at the specified time point post-Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 126 | 129
Percentage of participants | 85.7 [78.4 to 91.3] | 7.8 [3.8 to 13.8]

2. Secondary Outcome: Anti-gE Antibody Concentrations Expressed as Geometric Mean Concentrations (GMCs) and Between-group GMC Ratios
Description: Anti-gE antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as GMCs in milli-international units per milliliter (mIU/mL).
Time Frame: At 1 month post-Dose 2 of study intervention administration (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 126 | 129
mIU/mL | 26863.85 [20125.47 to 35858.35] | 1360.48 [1134.23 to 1631.85]
Statistical Analysis 1: Comparison: HZ/suSeq Group vs Placebo Group; To demonstrate the immunogenicity of HZ/su vaccine compared to Placebo, in terms of anti-gE GMCs, at 1 month post-Dose 2 of study intervention administration (Month 3); Test type: Superiority — The superiority was to be concluded if the lower limit (LL) of the 95% confidence interval (CI) of the adjusted GMC ratio between the HZ/su Group and Placebo Group for anti-gE antibody concentrations was equal to or above (>=) 3; ANOVA; GMC Ratio = 19.80, 95% CI 2-sided [14.09 to 27.82]

3. Secondary Outcome: Percentage of Participants Reporting Solicited Administration Site Events
Description: The assessed solicited administration site events included injection site erythema, pain, pruritus and swelling.
Time Frame: Within 7 days after each study intervention dose and across doses (vaccine/placebo administered at Day 1 and Month 2)
Population: This analysis was performed on the Exposed Set, which included all participants who received at least 1 dose of the study intervention and with the diary cards completed post-each study intervention dose.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants
  Erythema, post-Dose 1 | 0 [0 to 2.5] | 0 [0 to 2.5]
  Erythema, post-Dose 2: number analyzed (Participants) | 142 | 143
  Erythema, post-Dose 2 | 0.7 [0.0 to 3.9] | 0 [0 to 2.5]
  Erythema, Across doses | 0.7 [0 to 3.8] | 0 [0 to 2.5]
  Pain, post-Dose 1 | 53.1 [44.6 to 61.5] | 33.8 [26.2 to 42.1]
  Pain, post-Dose 2: number analyzed (Participants) | 142 | 143
  Pain, post-Dose 2 | 46.5 [38.1 to 55.0] | 37.8 [29.8 to 46.2]
  Pain, Across doses | 67.1 [58.8 to 74.8] | 49.0 [40.6 to 57.4]
  Pruritus, post-Dose 1 | 9.1 [4.9 to 15.0] | 8.3 [4.3 to 14.0]
  Pruritus, post-Dose 2: number analyzed (Participants) | 142 | 143
  Pruritus, post-Dose 2 | 12.7 [7.7 to 19.3] | 6.3 [2.9 to 11.6]
  Pruritus, Across doses | 20.3 [14.0 to 27.8] | 13.1 [8.1 to 19.7]
  Swelling, post-Dose 1 | 1.4 [0.2 to 5.0] | 0 [0 to 2.5]
  Swelling, post-Dose 2: number analyzed (Participants) | 142 | 143
  Swelling, post-Dose 2 | 0.7 [0.0 to 3.9] | 0 [0 to 2.5]
  Swelling, Across doses | 2.1 [0.4 to 6.0] | 0 [0 to 2.5]

4. Secondary Outcome: Percentage of Participants Reporting Solicited Systemic Events
Description: The assessed solicited systemic events included fatigue, fever, gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia and shivering.
Time Frame: Within 7 days after each study intervention dose and across doses (vaccine/placebo administered at Day 1 and Month 2)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants
  Fatigue, post-Dose 1 | 32.2 [24.6 to 40.5] | 15.2 [9.8 to 22.1]
  Fatigue, post-Dose 2: number analyzed (Participants) | 142 | 143
  Fatigue, post-Dose 2 | 35.2 [27.4 to 43.7] | 14.7 [9.3 to 21.6]
  Fatigue, Across doses | 44.8 [36.4 to 53.3] | 24.1 [17.4 to 31.9]
  Fever, post-Dose 1 | 26.6 [19.5 to 34.6] | 6.9 [3.4 to 12.3]
  Fever, post-Dose 2: number analyzed (Participants) | 142 | 143
  Fever, post-Dose 2 | 17.6 [11.7 to 24.9] | 3.5 [1.1 to 8.0]
  Fever, Across doses | 28.0 [20.8 to 36.1] | 9.7 [5.4 to 15.7]
  Gastrointestinal symptoms, post-Dose 1 | 4.2 [1.6 to 8.9] | 2.1 [0.4 to 5.9]
  Gastrointestinal symptoms, post-Dose 2: number analyzed (Participants) | 142 | 143
  Gastrointestinal symptoms, post-Dose 2 | 2.8 [0.8 to 7.1] | 0.7 [0.0 to 3.8]
  Gastrointestinal symptoms, Across doses | 7.0 [3.4 to 12.5] | 2.8 [0.8 to 6.9]
  Headache, post-Dose 1 | 16.1 [10.5 to 23.1] | 13.1 [8.1 to 19.7]
  Headache, post-Dose 2: number analyzed (Participants) | 142 | 143
  Headache, post-Dose 2 | 20.4 [14.1 to 28.0] | 11.9 [7.1 to 18.4]
  Headache, Across doses | 28.7 [21.4 to 36.8] | 22.8 [16.2 to 30.5]
  Myalgia, post-Dose 1 | 16.8 [11.1 to 23.9] | 2.8 [0.8 to 6.9]
  Myalgia, post-Dose 2: number analyzed (Participants) | 142 | 143
  Myalgia, post-Dose 2 | 13.4 [8.3 to 20.1] | 0.7 [0.0 to 3.8]
  Myalgia, Across doses | 22.4 [15.8 to 30.1] | 3.4 [1.1 to 7.9]
  Shivering, post-Dose 1 | 4.9 [2.0 to 9.8] | 4.1 [1.5 to 8.8]
  Shivering, post-Dose 2: number analyzed (Participants) | 142 | 143
  Shivering, post-Dose 2 | 4.9 [2.0 to 9.9] | 1.4 [0.2 to 5.0]
  Shivering, Across doses | 8.4 [4.4 to 14.2] | 5.5 [2.4 to 10.6]

5. Secondary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an AE that was not included in a list of solicited events using a participant diary. Unsolicited events must have been spontaneously communicated by a participant who had signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE.
Time Frame: Within 30 days after any study intervention dose administration (vaccine/placebo administered at Day 1 and Month 2)
Population: This analysis was performed on the Exposed Set, which included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants | 13.3 [8.2 to 20.0] | 13.1 [8.1 to 19.7]

6. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant or an abnormal pregnancy outcome, or an important medical event that may not have been life-threatening or resulted in death or hospitalization, but may have jeopardized the participant or required medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: From Dose 1 (Day 1) up to 30 days post-last study intervention dose
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants | 0.7 [0.0 to 3.8] | 0 [0 to 2.5]

7. Secondary Outcome: Percentage of Participants Reporting Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs were defined as a subset of AEs of special interest that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune etiology.
Time Frame: From Dose 1 (Day 1) up to 30 days post-last study intervention dose
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants | 0 [0 to 2.5] | 0 [0 to 2.5]

8. Secondary Outcome: Percentage of Participants Reporting SAEs
Description: as for outcome 6
Time Frame: From Dose 1 (Day 1) up to study end (Month 8)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants | 0.7 [0.0 to 3.8] | 1.4 [0.2 to 4.9]

9. Secondary Outcome: Percentage of Participants Reporting pIMDs
Description: as for outcome 7
Time Frame: From Dose 1 (Day 1) up to study end (Month 8)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 143 | 145
Percentage of participants | 0 [0 to 2.5] | 0 [0 to 2.5]

10. Secondary Outcome: Anti-gE Antibody Concentrations Expressed as GMCs
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At pre-study intervention administration (Day 1) and at 1 month post-Dose 2 of study intervention administration (Month 3)
Population: This analysis was performed on the Per Protocol Set, which included all eligible participants who received all doses as per protocol, complied with allowed dosing/blood draw intervals, without intercurrent conditions that may have interfered with immunogenicity, without prohibited concomitant medication/vaccination and with immunogenicity results available at the specified time points pre- and post-Dose 2.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 126 | 129
mIU/mL
  At Day 1 | 1210.86 [982.17 to 1492.79] | 1217.81 [1019.01 to 1455.39]
  At Month 3 | 26863.85 [20125.47 to 35858.35] | 1360.48 [1134.23 to 1631.85]

11. Secondary Outcome: Percentage of Participants Seropositive for Anti-gE Antibodies
Description: A participant seropositive for anti-gE antibodies was defined as a participant whose antibody concentration was greater than or equal to (>=) the assay cut-off value (97 mIU/mL).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 126 | 129
Percentage of participants
  At Day 1 | 97.6 [93.2 to 99.5] | 96.9 [92.3 to 99.1]
  At Month 3 | 99.2 [95.7 to 100.0] | 100 [97.2 to 100]

12. Secondary Outcome: Mean Geometric Increase (MGI) of Anti-gE Antibody Concentrations
Description: MGI was defined as the geometric mean of the within participant ratios of anti-gE antibody concentration at 1 month post-Dose 2 (Month 3) compared to pre-study intervention administration (Day 1) anti-gE antibody concentration.
Time Frame: At 1 month post-Dose 2 of study intervention administration (Month 3) compared to pre-study intervention administration (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | HZ/suSeq Group | Placebo Group
Number analyzed (Participants) | 126 | 129
Ratio | 22.19 [15.46 to 31.83] | 1.12 [0.92 to 1.36]

ADVERSE EVENTS:
Time Frame: Solicited administration site and systemic AEs: during the 7-day (Days 1-7) follow-up period after vaccination; Unsolicited AEs: during the 30-day (Days 1-30) follow-up period after vaccination; SAEs: from Dose 1 (Day 1) up to study end (Month 8).
Arm/Group | HZ/suSeq Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/145
Serious Adverse Events (participants affected / at risk) | 1/143 | 2/145
Other Adverse Events (participants affected / at risk) | 103/143 | 88/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/suSeq Group (N=143) | Placebo Group (N=145)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/suSeq Group (N=143) | Placebo Group (N=145)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (10) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Administration site erythema (General disorders) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 96 (142) | 71 (103)
Administration site swelling (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 12 (14) | 8 (8)
Fatigue (General disorders) | 64 (97) | 36 (46)
Pyrexia (General disorders) | 42 (65) | 16 (17)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 34 (45) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 42 (54) | 37 (43)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (31) | 19 (21)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT05219253/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT05219253/SAP_001.pdf